CLINICAL TRIAL: NCT04100798
Title: Clinical and Radiographic Evaluation of the Entire Papilla Preservation (EPP) Technique Versus Modified Minimally Invasive Surgical Technique (M-MIST) in Treatment of Intraosseous Defects in Patients With Stage III Periodontitis: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Ebrahim Mohamed Mokhtar, PHD Candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER 3-3-2
Record Dates: First submitted 2019-09-21; First posted 2019-09-24 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Intrabony Periodontal Defect

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Entire Papilla Preservation (EPP) technique (Experimental): A minimally invasive surgical technique that involves using a vertical incision away from the defect area in order to preserve the integrity of the related interdental papilla and elevating a full thickness flap then using microsurgical instruments to properly debride the intraosseous defect before closing the flap
  Interventions: Procedure: Entire Papilla Preservation technique
- Modified Minimally invasive Surgical Technique (M-MIST) (Active Comparator): A minimally invasive surgical technique that involves using a horizontal interdental incision that extends to the buccal aspect of the two teeth adjacent to the intraosseous defect then elevating a full thickness flap then using microsurgical instruments to properly debride the intraosseous defect before closing the flap
  Interventions: Procedure: Modified Minimally invasive Surgical Technique

INTERVENTIONS:
Procedure: Entire Papilla Preservation technique — A minimally invasive technique that allow access to the intrabony defect without affecting the interdental papilla related to it
  Other Names: EPP
  Arms: Entire Papilla Preservation (EPP) technique
Procedure: Modified Minimally invasive Surgical Technique — a minimally invasive technique that allow access to the intrabony defect area from the buccal aspect through a horizontal incision below the papilla without elevating it.
  Other Names: M-MIST
  Arms: Modified Minimally invasive Surgical Technique (M-MIST)

SUMMARY:
Periodontitis is defined as loss of periodontal attachment due to microbial associated host mediated inflammation. This would lead to the apical migration of the junctional epithelium allowing the bacterial biofilm to undergo apical widespread along the root surfaces of teeth causing bone resorption (Tonetti, Greenwell, & Kornman, 2018).

The main objective of periodontal surgeries is directed at complete preservation of the interdental soft tissues to achieve primary closure over the intraosseous defected sites during the early phases of wound healing. Evidence shows that surgical techniques are highly predictable in the treatment of pockets associated with deep and shallow intrabony defects affected majorly by the selected flap design. The purpose of the flap design of minimally invasive periodontal surgery is to overcome the drawbacks of conventional periodontal surgeries decreasing the surgical trauma, improving the clot stability, reducing patient discomfort post operatively and minimizing the surgical chair time (Aslan, Buduneli, & Cortellini, 2017b) Modified Minimally Invasive Surgical Technique (M-MIST) is considered one of the latest minimally invasive techniques that have been used in the treatment of intraosseous defects, this technique however entails an incision over the defect-associated interdental papilla that may jeopardize the volume and complex vascular integrity of the interdental tissues, lacking the special flap design that would emphasis clot stability for better wound healing. Where a new surgical technique turned entire papilla preservation has been developed for protection of the wound without affecting the vascularity of the area. (Pierpaolo Cortellini & Tonetti, 2015) This randomized clinical trial compared the clinical and radiographic efficacy of entire papilla preservation surgical technique (EPP) to Modified minimally invasive surgical technique (M-MIST) in the treatment of periodontal intraosseous defects in stage III periodontitis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 20 and 60 years old.
* Stage III periodontitis patient having 2 or 3 walled or combined 2 and 3 walled intraosseous defect ≥ 3 mm deep (assessed by trans-gingival probing, radiographic examination) with clinical attachment level (CAL) ≥ 5mm and pocket depth (PD) ≥ 6 mm.
* Defect not extending to a root furcation area.
* Vital teeth
* No history of intake of antibiotics or other medications affecting the periodontium in the previous 6 months.
* Patients who are cooperative, motivated, and hygiene conscious.

Exclusion Criteria:

* Any systemic disease that contra-indicates periodontal surgery or may affect healing.
* Smokers
* Pregnant females
* Drug abusers

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-08 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Clinical attachment Level gain (CAL gain) | 12 months
  CAL gain will be determined by measuring the distance from the cemento-enamel junction to the base of the pocket using a UNC 15 periodontal probe.

SECONDARY OUTCOMES:
Pocket depth (PD) | 12 months
  Probing depth will be measured from the gingival margin to the base of the periodontal pocket using a UNC 15 periodontal probe.
Gingival recession (GR) | 12 months
  Gingival recession will be measured using UNC periodontal probe from the cemento-enamel junction till the gingival margin (Ainamo & Bay, 1975).
Radiographic defect fil | 12 months
  The depth of intra-bony defect (IBD) will be measured from the alveolar bone crest to the base of the defect to detect the amount of bone fill Radiographs will be scanned and the radiographic IBD depth will be measured by a computer-aided software program
Gingival bleeding score | 12 months
  * Gingival bleeding score will be performed through gentle probing of the orifice of the gingival crevice from all four surfaces of all teeth using UNC Periodontal probe.
  * Recorded as (+) if bleeding is present or (-) if bleeding is absent.
  * If bleeding occurs within 10 seconds a positive finding is recorded and the number of positive sites is recorded and then expressed as a percentage of the number of sites examined
Post-surgical patient satisfaction | 12 months
  * Three questionnaires will be asked to determine patients' satisfaction with the outcome of surgery
  * Considering this was an elective operation, how likely would you be to recommend it to others?
  * If you had to make the decision again, how likely would you be to undergo this surgery'?
  * Considering everything, how satisfied are you with the outcome of your surgery
  * These questions could all be answered by the patient using a 7-point response scale where: Very Satisfied = 7; Not At All Satisfied = 1. (H. A. Kiyak et al., 1984)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided